CLINICAL TRIAL: NCT02260622
Title: A Phase 2, Open Label, Pilot Study to Examine the Use of Rivaroxaban Plus Aspirin vs. Clopidogrel Plus Aspirin for the Prevention of Restenosis After Infrainguinal Percutaneous Transluminal Angioplasty for Critical Limb Ischemia
Brief Title: Pilot Study to Examine the Use of Rivaroxaban After Angioplasty for Critical Limb Ischemia
Acronym: RIVAL-PAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20130484-01H
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Results first posted 2019-11-22 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-11

CONDITIONS: Critical Limb Ischemia
Keywords: Restenosis; Critical Limb Ischemia; Infrainguinal Percutaneous Transluminal Angioplasty; Rivaroxaban; Clopidogrel
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Rivaroxaban; Aspirin; Clopidogrel; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- clopidogrel plus aspirin (Active Comparator): Clopidogrel 75 mg daily X 90 days plus ASA 81 mg daily
  Interventions: Drug: clopidogrel plus aspirin
- rivaroxaban plus aspirin (Experimental): Rivaroxaban 2.5 mg BID X 90 days plus ASA 81 mg daily
  Interventions: Drug: rivaroxaban plus aspirin

INTERVENTIONS:
Drug: rivaroxaban plus aspirin — Rivaroxaban 2.5 mg twice daily for 90 days (rivaroxaban will be started 6 to 8 hours after the finalization of the procedure) and 81 mg of ASA daily for 90 days
  Other Names: treatment arm
  Arms: rivaroxaban plus aspirin
Drug: clopidogrel plus aspirin — Clopidogrel 75 mg daily for 90 days (with a loading dose of 300 mg clopidogrel following PTA) and 81 mg of ASA daily for 90 days
  Other Names: Plavix plus ASA; Standard Care
  Arms: clopidogrel plus aspirin

SUMMARY:
Background: Up to 10% of patients with peripheral arterial disease (PAD) will develop critical limb ischemia (CLI) which is a decrease of blood flow in the arteries of the limb. CLI results in resting pain, ulcers, gangrene, and limb loss. The outcome for patients with CLI is poor. Within 3 months of onset, 12% of patients will require an amputation (removal of part of the limb) and 9% will die of major cardiovascular events (heart attack or stroke). Percutaneous angioplasty (PTA), a procedure used to open the blockages in blood flow, has become the first-line treatment for CLI given its effectiveness, lower cost, and lower risk of complications. However, 40% of patients will have re-narrowing of the arteries (restenosis) following the PTA procedure. This is thought to happen in part due to build up of blood cells called platelets which can also lead to the formation of blood clots. In order to try to avoid this problem, most patients are prescribed a combination of two blood thinning medications, acetylsalicylic acid (ASA or aspirin) and clopidogrel (the brand name is Plavix).

The purpose of this study is to determine if a new blood thinner called rivaroxaban, given in combination with aspirin, would be more effective in preventing re-narrowing of the arteries than the current standard of care (aspirin and clopidogrel).

Rivaroxaban is a pill and does not require blood test monitoring. It has been approved by Health Canada for use in prevention of blood clots in patients undergoing hip or knee surgery and to treat patients with blood clots in their legs and lungs. Low dose aspirin has been approved for reducing the risk of heart attacks and strokes. These medications have not been tested together in patients for prevention of re-narrowing of their arteries

This is a pilot study conducted at one center, The Ottawa Hospital.

It is a Phase 2 open label randomized controlled trial.

Following the PTA procedure, once all inclusion/exclusion criteria are met, the participant will be randomized into one of two groups:

1. Rivaroxaban 2.5 mg BID X 90 days plus ASA 81 mg daily OR
2. Clopidogrel 75 mg daily X 90 days plus ASA 81 mg daily

Visits will occur at 7 days, 30 days, 90 days, 6 months and 12 months. Participants will be followed for 12 months (± 14 days) in total. All adverse events will be collected for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Infra-inguinal PAD presenting as CLI defined as a Rutherford category of 3, 4, or 5
3. More than 50% stenosis in the target infrainguinal vessel
4. Good candidates for PTA using POBA (plain old balloon angioplasty) with or without stenting defined as TASC a and b lesions.

Exclusion Criteria:

1. Rutherford scale of 0,1,2 or 6
2. Acute limb-threatening ischemia (e.g. embolic disease)
3. Previous infrainguinal bypass or PTA procedures of the affected leg
4. Hybrid procedures
5. Creatinine clearance <30 mL/min
6. Platelet count <100x109/L
7. INR >1.5; Hbg <100 g/L
8. History of or condition associated with increased bleeding risk including, but not limited to:

   1. Major surgical procedure or trauma within 30 days before the randomization visit
   2. Clinically significant gastrointestinal bleeding within 6 months before the randomization visit
   3. History of intracranial, intraocular, spinal, or atraumatic intra-articular bleeding
   4. Chronic hemorrhagic disorder
   5. Known intracranial neoplasm, arteriovenous malformation, or aneurysm
   6. Sustained uncontrolled hypertension: systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥100 mmHg
9. Severe, disabling stroke (modified Rankin score of 4 to 5, inclusive) within 3 months or any stroke within 14 days before the randomization visit
10. Aspirin in combination with thienopyridines within 5 days before randomization
11. Intravenous antiplatelets within 5 days before randomization
12. Fibrinolytics within 10 days before randomization
13. Known HIV infection at time of screening
14. Known significant liver disease (e.g., acute clinical hepatitis, chronic active hepatitis, cirrhosis or ALT >3ULN)
15. Childbearing potential without proper contraceptive measures, pregnancy or breast feeding
16. Drug addiction or alcohol abuse within 12 months before the randomization visit
17. Systemic treatment with strong CYP 3A4 and P-glycoprotein inhibitors : such as ketoconazole, itraconazole, posaconazole, or ritonavir
18. Known allergy or hypersensitivity to any component of rivaroxaban, ASA or clopidogrel
19. Need for long term anticoagulation or double antiplatelet agents other than PAD such as atrial fibrillation, heart valve replacement, acute coronary syndrome, stroke or venous thromboembolism
20. Anticipated need for chronic (> 4 weeks) therapy with non-steroidal anti-inflammatory drugs.
21. Concomitant treatment with any other anticoagulant, including oral anticoagulants, such as warfarin, dabigatran, apixaban, except under circumstances of switching therapy to or from study treatment.
22. Inability to adhere to protocol.
23. Severe concomitant condition or disease (e.g. life expectancy <6 months secondary to cancer, advanced liver disease or dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10; Primary Completion 2017-06 (Actual); Study Completion 2019-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Gandara, MD, Principal Investigator — Ottawa Hospital Research Institute; Prasad Jetty, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Started | 11 | 9
Completed | 11 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin | Total
Number analyzed (Participants) | 11 | 9 | 20
Age, Continuous [Mean (Full Range); unit: years] | 74.8 [55 to 84] | 59.5 [54 to 82] | 67 [54 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 7 | 5 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 8 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Reintervention, Above Ankle Amputation and Restenosis (RAS)
Description: The primary outcome is a combined endpoint consisting of any Reintervention (surgical procedures to revascularize), Above ankle amputation and restenosis(recurrence of blockage in the vein) (RAS) at one year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Number analyzed (Participants) | 11 | 9
Participants | 7 | 4

2. Secondary Outcome: Number of Participants With 2 Class Improvement on the Rutherford Scale
Description: Clinical improvement defined as cumulative improvement of 2 classes of the Rutherford scale without the need for repeated TLR in surviving patients.
  There are seven stages to consider. the lower the score the less severe the disease or condition.
  Rutherford Scale:
  Stage 0 - Asymptomatic Stage 1 - Mild claudication Stage 2 - Moderate claudication - The distance that delineates mild, moderate and severe claudication is not specified in the Rutherford classification, but is mentioned in the Fontaine classification as 200 meters.
  Stage 3 - Severe claudication Stage 4 - Rest pain Stage 5 - Ischemic ulceration not exceeding ulcer of the digits of the foot Stage 6 - Severe ischemic ulcers or frank gangrene
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Number analyzed (Participants) | 11 | 9
Participants | 5 | 8

3. Secondary Outcome: Event-free Survival
Description: Event-free survival How long a patient is alive without the need for any further intervention or vascular events.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Number analyzed (Participants) | 11 | 9
Participants | 4 | 4

4. Secondary Outcome: Overall Survival
Description: Overall survival. How long a patient is alive following the intervention.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Number analyzed (Participants) | 11 | 9
Participants | 11 | 9

5. Secondary Outcome: The Number of Patients Requiring Target Lesions Revascularization Between Day 1 and the Final Visit (TLR)
Description: Target lesion revascularization (TLR) between day 1 and final visit
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Number analyzed (Participants) | 11 | 9
Participants | 2 | 1

6. Secondary Outcome: TVR
Description: Target vessel revascularization (TVR between day 1 and final visit)
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Number analyzed (Participants) | 11 | 9
Participants | 2 | 1

7. Secondary Outcome: Peri-procedure Death
Description: The number of patients that die within 30 days of the revascularization procedure.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Number analyzed (Participants) | 11 | 9
Participants | 0 | 0

8. Secondary Outcome: MACE
Description: Cumulative rate of major adverse cardiovascular events between day 1 and final visit
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Number analyzed (Participants) | 11 | 9
Participants | 0 | 0

9. Secondary Outcome: Major Bleeding
Description: Cumulative rate of major bleeding between day 1 and day 90
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Number analyzed (Participants) | 11 | 9
Participants | 0 | 0

10. Secondary Outcome: Minor Bleeding
Description: Cumulative clinically relevant or minor bleeding between day 1 and day 90
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Number analyzed (Participants) | 11 | 9
Participants | 0 | 1

11. Secondary Outcome: Biomarkers
Description: Biological plausibility by measuring coagulation changes and SMC proliferation markers within 7 and 90 days based on the following markers: D-dimer, soluble CD40/44 ligands, and ERK 1/2
Time Frame: 90 days
Population: Not performed.
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: From randomization to 12-month follow-up
Arm/Group | Clopidogrel Plus Aspirin | Rivaroxaban Plus Aspirin
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/9
Other Adverse Events (participants affected / at risk) | 2/11 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel Plus Aspirin (N=11) | Rivaroxaban Plus Aspirin (N=9)
Leg injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Abnormal Lab Result (Investigations) | 1 (1) | 0 (0)
Minor Bleed - not clinically relevant (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-04): https://cdn.clinicaltrials.gov/large-docs/22/NCT02260622/Prot_SAP_000.pdf